CLINICAL TRIAL: NCT06935981
Title: The Effect of School-Based Mental Health Program on Positive Mental Health and Self-Esteem Levels in Adolescents
Brief Title: Effectiveness of School-based Mental Health Program
Acronym: ADOLESCENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Lok (Other)
Responsible Party: Sponsor-Investigator, Neslihan Lok, PROF. DR., Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SelçukU-ZAYDIN-001; 23212017 (Other Grant/Funding Number: SELCUK UNIVERSITY)
Record Dates: First submitted 2025-04-05; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Adolescent; Mental Health; Mental Health Care; Mental Health Conditions
Keywords: Positive mental health; Self-confidence; Mental health program; Adolescence; Psychiatric nursing
MeSH Terms: conditions — Psychological Well-Being | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: This study protocol describes a randomized controlled trial with a parallel group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Nursing interventions will last 8 weeks and consist of education, counseling and homework.
  Interventions: Other: school-based mental health program
- control group (No Intervention): No intervention will be performed and 8 weeks of nursing interventions will be applied after the final tests are collected.

INTERVENTIONS:
Other: school-based mental health program — Week 1 Session 1-Beginning-Getting Acquainted Week 2 Session 2-Emotion, Thought and Behavior Wheel Week 3 Session 3- Optimism Week 4 Session 4- Forgiveness Week 5 Session 5- Saying No Week 6 Session 6- Effective Communication Week 7 Session 7- Problem Solving Week 8 Session 8- Saying Goodbye
  Other Names: guidance
  Arms: intervention group

SUMMARY:
Aim: This article presents the planned protocol for a study investigating the effects of an eight-week nursing intervention to be implemented in school on positive mental health and self-confidence levels of adolescents.

Design: This study protocol describes a randomized controlled trial with a parallel group design.

Method: Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Statement 2013 checklist is used in this study. The CONSORT (Consolidated Standards of Reporting Trials) flowchart is used in this protocol. The research population consists of 310 students studying in the 9th grade at Erbil Koru Anatolian High School located in Selçuklu district of Konya province. A total of 66 students were determined as intervention (33) and control (33) who met the inclusion and exclusion criteria. Nursing interventions will last for 8 weeks and consist of education, counseling and homework.

Conclusion: The results obtained from this study may help protect and develop the mental health of adolescents and guide future mental health programs.

DETAILED DESCRIPTION:
Purpose of the Study

The purpose of this study was to investigate the effects of an eight-week nursing intervention implemented in school on positive mental health and self-esteem. The specific objectives were as follows:

* to analyze the effectiveness of the intervention (education and counseling, and psychoeducation of nursing practices) in increasing positive mental health.
* to evaluate the feasibility of the intervention. Hypotheses H1: The positive mental health level of the intervention group receiving the School-Based Mental Health Program is higher than the control group.

H2: The self-esteem level of the intervention group receiving the School-Based Mental Health Program is higher than the control group.

Method The study is a randomized controlled trial with a parallel group design. It was prepared based on the Standard Protocol Items: Recommendations for Interventional Trials (Chan et al., 2013) and complies with the Consolidation Standards of Reporting Trials (CONSORT) statement (Moher et al., 2012).

Inclusion Criteria:

* 9th grade students who agree to participate in the study
* Those who score 78 or below on the Positive Mental Health Scale
* Those who score 3.5 or below on the Self-Confidence Level Scale

Exclusion Criteria:

* Those who have any mental illness,
* Those who participate in a similar program.

Exclusion Criteria:

* Those who do not attend at least 2 educational program sessions,
* The student or parent wants to leave the sessions. Randomization Students will be randomly assigned to the intervention and control groups. In order to reduce selection bias and control variables that may have an effect on the outcome variables, participants will be assigned to the experimental and control groups using the simple randomization method by a statistician other than the researcher. The intervention and control group sets will be created using the research randomizer computer program (www.randomizer.org). It will be ensured that the study complies with the inclusion-exclusion criteria and that each group consists of 33 students . Post-tests will be administered by an interviewer to avoid bias.

Outcome Measurements The results of the study will consist of positive mental health level (primary outcome) and self-confidence level (secondary outcome). Data will be collected using Participant Information Form, Personal Information Form, Positive Mental Health Scale and Self-Confidence Scale.

Personal Information Form A data form consisting of 10 questions based on literature and sociodemographic characteristics (age, gender, perceived health status, parental education status, parental attitude, perceived income level, school liking, participation in social activities, chronic mental illness status) prepared by the researcher.

Positive Mental Health Scale Positive mental health, defined as the presence of general emotional, psychological and social well-being, is an important factor of general mental health. It was developed by Lluch (1999) in order to define the concept of positive mental health and to evaluate the level of positive mental health. Its validity and reliability in Turkish were performed by Teke and Baysan Arabacı (2018). The four-point Likert-type scale, consisting of thirty-nine statements and six subgroups, has direct and reverse items. The sub-dimensions of the scale are; personal satisfaction (self-esteem, positive outlook on the future) (4, 6, 7, 12, 14, 31, 38, 39), prosocial attitude (altruistic social attitude, acceptance of different social characteristics) (1, 3, 23, 25, 37), self-control (skills for effectively coping with crisis and stress situations) (2, 5, 21, 22, 26), autonomy (ability to control one's behavior) (10, 13, 19, 33, 34), problem solving and self-actualization (developed decision-making abilities) (15, 16, 17, 27, 28, 29, 32, 35, 36), interpersonal relationship skills (empathy, understanding emotions) (8, 9, 11, 18, 20, 24, 30). Each item of the scale receives a score ranging from "4" to "1" for "always or almost always," "often," "sometimes," and "never or rarely," respectively. Statements 1, 2, 3, 6, 7, 8, 9, 10, 12, 13, 14, 19, 24, 30, 31, 33, 34, 38, and 39 are reverse statements and their scores are reversed. The scores to be obtained from the scale range from 39 to 156. High scores to be obtained from the scale indicate a high level of positive mental health. In the Turkish validity and reliability study, the Cronbach Alpha coefficient for the whole was found to be 0.93 and the Cronbach Alpha coefficients for the subscales were found to be αKM=0.80, αPT=0.86, αÖD=0.78, αÖ=0.86, αPÇKG=0.80 and αKIB=0.83 (Lluch, 1999; Teke and Baysan Arabacı, 2018).

Self-Confidence Scale The Self-Confidence Scale developed by Akın (2007) was used to assess the self-confidence levels of adolescents. The scale includes a 5-choice rating consisting of 33 items and two sub-dimensions as internal self-confidence and external self-confidence. There is no reverse item in the scale. The highest score that can be obtained from this scale is 165, and the lowest score is 33. The scale has two sub-dimensions as internal self-confidence and external self-confidence. It consists of items such as internal self-confidence (1, 3, 4, 5, 7, 9, 10, 12, 15, 17, 19, 21, 23, 25, 27, 30, 32) and external self-confidence (2, 6, 8, 11, 13, 14, 16, 18, 20, 22, 24, 26, 28, 29, 31, 33). By dividing the total score obtained from the scale by the number of items (33), a conclusion can be reached about the self-confidence level of the individual. A score below 2.5 on the Self-Confidence Scale indicates low, between 2.5 and 3.5 indicates medium, and 3.5 and above indicates high self-confidence. The Cronbach's alpha coefficients of the self-confidence scale for the whole scale are; 0.83, and 0.83 and 0.85 for the internal self-confidence and external self-confidence subscales, respectively (Akın, 2007).

Dependent Variables

* Positive Mental Health Scale Mean Score
* Self-Confidence Scale Mean Score

Independent Variables

* School-Based Mental Health Development Program Control Variables
* Sociodemographic characteristics (age, gender, parental education status of students) Study Procedure This study is a randomized controlled trial consisting of two groups, one intervention group and one control group. Adolescents in the intervention group will be provided with group education, counseling service, and homework assignments, and homework assignments will be used as reminders after the education. No intervention will be applied to the participants in the control group. Pretests and approval for participation in the study will be completed by the researchers before randomization, and posttests will be completed by the interviewer after the psychoeducation is completed. The study will last 8 weeks. Intervention Group: Education, counseling and homework will be applied to the intervention group. Post-tests will be applied at the end of week 8. Control Group: No intervention will be applied to the control group and post-tests will be applied at the end of week 8. After the post-tests are completed, the mental health education given to the intervention group will also be given to the control group.

Intervention and Time Content School-Based Mental Health Program's Topics Week 1 Session 1-Beginning-Getting Acquainted Week 2 Session 2-Emotion, Thought and Behavior Wheel Week 3 Session 3- Optimism Week 4 Session 4- Forgiveness Week 5 Session 5- Saying No Week 6 Session 6- Effective Communication Week 7 Session 7- Problem Solving Week 8 Session 8- Saying Goodbye

ELIGIBILITY:
Inclusion Criteria:

* • 9th grade students who agreed to participate in the study

  * Those who scored 78 and below on the Positive Mental Health Scale
  * Those who scored 3.5 and below on the Self-Confidence Level Scale

Exclusion Criteria:

* • Those who have any mental illness,

  * Those who participate in a similar program.

Ages: 14 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Positive Mental Health Scale | From enrollment to the end of training at 8 weeks
  Positive mental health, defined as the presence of general emotional, psychological and social well-being, is an important factor of general mental health. It was developed by Lluch (1999) in order to define the concept of positive mental health and to evaluate the level of positive mental health. Its validity and reliability in Turkish were performed by Teke and Baysan Arabacı (2018). The four-point Likert-format scale consisting of thirty-nine statements and six subgroups has reverse and direct items. The sub-dimensions of the scale are; personal satisfaction (self-esteem, positive outlook on the future) (4, 6, 7, 12, 14, 31, 38, 39), prosocial attitude (altruistic social attitude, acceptance of different social characteristics) (1, 3, 23, 25, 37), self-control (skills for effectively coping with crisis and stress situations) (2, 5, 21, 22, 26), autonomy (ability to control one's behavior) (10, 13, 19, 33, 34), problem solving and self-actualization (developed decision-making abilit
Self confidence scale | From enrollment to the end of training at 8 weeks
  In order to assess the self-confidence levels of adolescents, the Self-Confidence Scale developed by Akın (2007) was used. The scale includes 33 items and a 5-option rating consisting of two subdimensions as internal self-confidence and external self-confidence. There are no reverse items in the scale. The highest score that can be obtained from this scale is 165, and the lowest score is 33. The scale has two subdimensions as internal self-confidence and external self-confidence. It consists of items internal self-confidence (1, 3, 4, 5, 7, 9, 10, 12, 15, 17, 19, 21, 23, 25, 27, 30, 32) and external self-confidence (2, 6, 8, 11, 13, 14, 16, 18, 20, 22, 24, 26, 28, 29, 31, 33). By dividing the total score from the scale by the number of items (33), a conclusion can be reached about the individual's self-confidence level. A score below 2.5 indicates low self-confidence, between 2.5 and 3.5 indicates medium self-confidence, and 3.5 and above indicates high self-confidence. The Cronbach a

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Lök, Prof. Dr., Study Director — Selcuk University
Locations (1):
- Erbil Koru Anadolu Lisesi, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No